CLINICAL TRIAL: NCT03654196
Title: A Multicenter, Randomized, Double-blinded, Active-controlled, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of HL301 Versus Umkamin Tab. in Acute Bronchitis Patients
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of HL301 Versus Umkamin Tab in Acute Bronchitis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HL_HL301_301
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Acute Bronchitis
Keywords: Acute Bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HL301(Experimental) (Experimental): Total 7 days of treatment and The daily dose is as follows [Morning: HL301 1Tab + Placebo of Umkamin 1Tab] [Noon: Placebo of Umkamin 1Tab] [Evening: HL301 1Tab + Placebo of Umkamin 1Tab]
  Interventions: Drug: HL301(Experimental)
- Umkamin(Active Comparator) (Active Comparator): Total 7 days of treatment and The daily dose is as follows [Morning: Placebo of HL301 1Tab + Umkamin 1Tab] [Noon: Umkamin 1Tab] [Evening: Placebo of HL301 1Tab + Umkamin 1Tab]
  Interventions: Drug: Umkamin(Active Comparator)

INTERVENTIONS:
Drug: HL301(Experimental) — Total 7 days of treatment and The daily dose is as follows [Morning: HL301 1Tab + Placebo of Umkamin 1Tab] [Noon: Placebo of Umkamin 1Tab] [Evening: HL301 1Tab + Placebo of Umkamin 1Tab]
  Other Names: HL301 and Placebo of Umkamin
  Arms: HL301(Experimental)
Drug: Umkamin(Active Comparator) — Total 7 days of treatment and The daily dose is as follows [Morning: Placebo of HL301 1Tab + Umkamin 1Tab] [Noon: Umkamin 1Tab] [Evening: Placebo of HL301 1Tab + Umkamin 1Tab]
  Other Names: Placebo of HL301 and Umkamin
  Arms: Umkamin(Active Comparator)

SUMMARY:
A Multicenter, Randomized, Double-blinded, Active-controlled, Parallel, Phase III Clinical Trial to Evaluate the Efficacy and Safety of HL301 versus Umkamin tab. in acute bronchitis patients

Endpoint: BSS, The improvement and improvement rate of the tester for the treatment response, The satisfaction of the subject

ELIGIBILITY:
Inclusion Criteria:

1. Both gender, 19 years ≤ age ≤ 80 years
2. (Bronchitis Severity Score)* ≥ 5point at Visit 2 (Randomized Visit)
3. Acute bronchitis within 48hr based on Visit 2 (Randomized Visit)
4. Those who can comply with the requirements of clinical trials
5. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. Patients with respiratory and systemic infections requiring systemic antibiotic therapy
2. Patients with bleeding tendency
3. Patients who investigators determines to severe respiratory disease that would interfere with study assessment
4. Patients who were treated with oral systemic adrenocortical hormone or immunosuppressive drug within 4 weeks prior to Visit 2
5. Patients who were treated with oral antihistamines, ACE suppressive. or systemic/inhalative glucocorticosteroid within 2 weeks prior to Visit 2

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Bronchitis Severity Total Score(BSS) Change | Visit 1 (-3 day), Visit 2 (0 day), Visit 3 (7 day)
  The BSS comprises the following five symptoms typical for Acute Bronchitis: cough, sputum, rales on auscultation, chest pain on coughing, and dyspnoea. These symptoms are each assessed according to a 5-point Likert scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe

SECONDARY OUTCOMES:
The improvement and improvement rate of the tester for the treatment | Visit 3 (7 day)
  Improvement and improvement rate are assessed by tester according to a 5 factors: Deterioration, No change, Slight to moderate improvement, Major improvement, Complete recovery
The satisfaction of the subject (Questionnaire) | Visit 3 (7 day)
  Satisfaction of the subject (Questionnaire) are assessed by subject according to a 5 factors: Very dissatisfied, Dissatisfied, Neutral, Satisfied, Very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Hospital, Seoul, Dongdaemun-gu, South Korea